CLINICAL TRIAL: NCT03067636
Title: Retraining the Body and Brain to Conquer Compulsions
Brief Title: Retraining Body and Brain to Conquer Compulsions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Rebecca Segrave, Dr Rebecca Segrave, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160437
Record Dates: First submitted 2017-02-23; First posted 2017-03-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Compulsive Behavior
MeSH Terms: conditions — Compulsive Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical exercise + stress management activity A (Active Comparator): Eight week program of concurrent exercise and stress management training.
  Interventions: Behavioral: Physical Exercise; Behavioral: Stress management training A
- Physical exercise + stress management activity B (Active Comparator): Eight week program of concurrent exercise and stress management training.
  Interventions: Behavioral: Physical Exercise; Behavioral: Stress management training B
- Lifestyle as usual (No Intervention): Eight weeks period with no alteration of usual lifestyle.
  Participants randomized to this arm are eligible for re-randomisation to one of the active conditions at the conclusion of week eight.

INTERVENTIONS:
Behavioral: Physical Exercise — Physical exercise: Amount of time exercising gradually titrated from 90-minutes in week one to 180-minutes in week eight. Intensity titrated concurrently from 40 - 60% VO2 max in week one to 40 - 90% VO2 max in week eight. Eight week gym membership provided to all participants to facilitate engagement in exercise.
  Arms: Physical exercise + stress management activity A; Physical exercise + stress management activity B
Behavioral: Stress management training A — Stress management training A: Daily stress management training for eight weeks with training activity delivered via app. Session lengths titrated from 10-minutes per day in the first week to 20-minutes per day in week eight.
  Arms: Physical exercise + stress management activity A
Behavioral: Stress management training B — Stress management training B: Daily stress management training for eight weeks with training activity delivered via app. Session lengths titrated from 10-minutes per day in the first week to 20-minutes per day in week eight.
  Arms: Physical exercise + stress management activity B

SUMMARY:
Following the realisation that many aspects of the way we live our life, such as our diet, activity levels, and amount of screen time, can have a potent impact on mental health and brain functioning 'lifestyle' based interventions have become topical in medical research. In particular, much scientific attention has been devoted to the impact of physical exercise and various stress reduction techniques on mood disorders. We aim to extend this work and investigate their impact on compulsivity.

We will do this by conducting a pilot proof-of-principal intervention study. The study will compare the impact of eight-weeks of:

1. regular physical exercise + stress management activity A,
2. regular physical exercise + stress management activity B,
3. lifestyle as usual.

The participant cohort will be adults who endorse mild-moderate behavioural compulsivity on one of the following domains:

* drinking alcohol
* gambling
* eating
* washing or cleaning
* checking
* ordering or arranging objects

DETAILED DESCRIPTION:
This study is investigating the impact of regular physical exercise and stress management activities on mental health and brain function. It is specifically focusing on how engaging in these activities might impact activity in brain circuits associated with compulsivity, and help to reduce compulsive patterns of behaviour.

A compulsive behaviour is something that we do regularly, feel pressured to do, and have difficulty stopping even though it is not benefiting us. Having compulsive patterns of behaviour is very common. It's been estimated that as many as 80% of the general population experience compulsivity at some point in their lives. That's most of us! Compulsive behaviours range in severity from mild to entrenched, and can take many forms. For example, gambling too often or washing ones hands excessively. For some people what starts out as a mild pattern of behaviour, such as a glass of wine every night after a stressful day, can develop into a problem, like alcohol dependence. As so many people experience mild to moderate compulsivity it would be helpful to have accessible evidence-based strategies that reduce compulsive tendencies.

One promising candidate is physical exercise. In addition to the well-known physical health benefits, regular exercise also has a potent positive effect on brain health and mental well being. Other candidates are specific stress management activities. Certain stress management techniques, such as brain training, meditation, psycho-education, music therapy, yoga, and guided relaxation, can promote optimal mental health, improve cognitive functioning and help keep the body's physiological arousal systems within a healthy range. Some stress management activities may also help to reduce compulsive behavioural patterns. Importantly, as physical exercise increases neuroplasticity (i.e. malleability of the brain), engaging in regular exercise may enhance the effectiveness of concurrent stress management activities.

This research study is investigating the impact of eight-weeks of regular physical exercise paired with two different stress management activities on brain health, mental health, and compulsivity. Both of these activities have previously been shown to reduce stress and improve mental health, we are investigating whether one is more effective than the other.

As regular exercise and stress management training are time consuming, taking part in the study will reduce the opportunity to engage in compulsive behaviours. As such, our primary focus for the study will not be a reduction in the time spent engaging in compulsive behaviour. Instead, we will focus on whether the interventions modulate aspects of brain function associated with compulsivity (e.g. hippocampal integrity, functional brain activity during reward processing), aspects of cognition associated with compulsivity (e.g. affective processing bias and decision making), indices of the bodies stress system (e.g. cortisol awakening response), and aspects of mental health and quality of life that can be compromised in sub-clinical compulsive populations (e.g. experiential avoidance, general well being, symptoms of anxiety and depression).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to provide informed consent,
* Endorse current behavioural compulsiveness in one of the following domains: alcohol consumption, gambling, eating, checking, washing/cleaning, ordering/arranging,
* Severity of compulsivity falls within mild-moderate range on transdiagnostic YBOCS,
* Level of physical activity fell within WHO Global Recommendations on Physical Activity for Health guidelines definitions of 'sedentary/inactive' across the prior three months, and for a minimum of four of the prior six months.
* Ability to adhere to study procedures.

Exclusion Criteria:

* Lifetime history of DSM-5 defined psychotic illness, severe substance use disorder, severe gambling disorder, binge eating disorder, bulimia nervosa,
* Current major depressive episode or anxiety disorder,
* History of neurological illness or moderate - severe brain injury,
* Have a major unstable medical illness or a chronic pain condition,
* Have a history of cardiovascular disease or musculoskeletal injury or disease that would preclude safe engagement in VO2 max testing or regular physical exercise,
* Lifetime diagnosis of learning difficulty, ADHD, other condition involving cognitive impairment as a primary feature,
* Severe claustrophobia, metallic implant within the body or other contraindication to MRI scanning,
* Shift work employment schedule within the prior 6-months,
* Endocrine disorder, adrenal dysfunction, autoimmune disorder, or other condition known to have a direct effect on the HPA axis,
* Psychoactive or glucocorticoid medications within the past month,
* Currently pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change in hippocampal integrity | Baseline (0 months), post (2 months)
  Composite score of hippocampal health indices, including volume (structural MRI) and neuronal NAA levels (MRS).

SECONDARY OUTCOMES:
Change in functional activation during reward processing | Baseline (0 months), post (2 months)
  fMRI Monetary Incentive Delay Task
Change in cortisol awakening reponse | Baseline (0 months), post (2 months), follow up (three months)
  Salivary cortisol
Change in affective processing bias | Baseline (0 months), post (2 months), follow up (three months)
  BeanFest
Change in risky decision making | Baseline (0 months), post (2 months), follow up (three months)
  Balloon Analogue Risk Task
Change in behavioral compulsivity | Baseline (0 months), post (2 months), follow up (three months)
  Transdiagnositc YBOCS
Change in psychosocial well being | Baseline (0 months), post (2 months), follow up (three months)
  Battery of self-report mental health and well being questionnaires assessing: symptoms of depression and anxiety, experiential avoidance, tolerance of uncertainly, impulsivity, obsession beliefs, well being, self efficacy, quality of life, and quality of inter-personal support.
Change in physical fitness | Baseline (0 months), post (2 months), follow up (three months)
  VO2 max

CONTACTS AND LOCATIONS:
Locations (1):
- Monash University, Brain and Mental Health Lab, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No